CLINICAL TRIAL: NCT01993342
Title: Determination of Adipocytokine in Synovial Fluid of Osteoarthritis Patients With Joint Pain and Effusion
Brief Title: Determination of Adipocytokine in Synovial Fluid of Osteoarthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, Joan Calvet Fontova, Dr, Parc Taulí Hospital Universitari
Other Study IDs: Joan03
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis
Keywords: adipocytokines; osteoarthritis; inflammation; ultrasonography
MeSH Terms: conditions — Osteoarthritis; Inflammation | interventions — Arthrocentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Synovial fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inflammatory knee osteoarthritis: We recruited patients with osteoarthritis and synovial effusion to diagnostic the effusion and to confirm that this this synovial fluid had mechanical characteristics. Now we are going to determine the adipocytokines and traditional parameters of inflammation in this synovial fluid to correlate it, and we will associate it with the ultrasound explanation of the knee that we have in our database.
  Interventions: Other: arthrocentesis; Other: ultrasonography of the knee

INTERVENTIONS:
Other: arthrocentesis — The made a diagnostic arthrocentesis to all patient we included
Other: ultrasonography of the knee — We explored the affected knee with an ultrasound explanation in order to describe inflammatory changes based on standard examination.

SUMMARY:
The purpose of this study is to determine the concentration of different adipocytokine (adiponectin, leptin, resistin, visfatin, osteopontin) and an inflammation classic markers as Interleukine 1 beta, tumor necrosis alfa, interleukine 6 and high sensibility reactive c protein in the synovial fluid of knee osteoarthritis patients, and compare with the inflammation detected with ultrasonography evaluation of the joint. In last years, some studies appeared focusing on the role of adipocytokines in osteoarthritis and they correlated adipocytokines with cartilage degradation and x-ray degree; in our study we will focused in the importance of adipocytokines in the inflammatory changes more than in joint destruction.

ELIGIBILITY:
Inclusion Criteria:

* aged 50 to 81
* primary osteoarthritis of the knee
* synovial effusion in examination
* patient who have the results in our database

Exclusion Criteria:

* any other rheumatic conditions as rheumatoid arthritis or another inflammatory disease
* secondary knee osteoarthritis
* history of knee surgery
* any conditions that at investigator criteria exclude the patient from study procedures

Ages: 50 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with knee osteoarthritis and synovial effusion who attende to a Rheumatologist unit for this problem. We made the visit and anonimously we kept the results of examination and ultrasonography in our database and we freezed synovial fluid. Now we will determine the adipocytokines and classic inflammatory parameters in this synovial fluid
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-11 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Determination of adipocytokine levels (adiponectin, leptin, resistin, visfatin, osteopontin) in synovial fluid | We determine adipocytoquines in one month, all patients in the same determination kit
  We have all the synovial fluid freeze, so now we have to determine the levels of everyone.

SECONDARY OUTCOMES:
Knee inflammation parameters detected by ultrasonography | three months
  We performed the ultrasonography evaluation at the same time than the visit were realized, and we have the results in a data base, so we will wait for the adipocytokine results and we will compare with ultrasound evaluation
To determine additional classic parameters of inflammation in synovial fluid as Interleukine 1 beta, Interleukine 6 and tumor necrosis factor alfa | We determine this inflammatory parameters in one month in all patient at the same time
  We will use classic inflammation parameters to compare with adipocytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Joan Calvet, Dr, Principal Investigator — Hospital Parc Tauli; Cristobal Orellana, Dr, Study Director — Hospital Parc Tauli
Locations (1):
- Hospital Parc Tauli Sabadell, Sabadell, Barcelona, Spain